CLINICAL TRIAL: NCT01581333
Title: Randomized Open Label Clinical Trial Directed to Optimize the Duration of Empirical Antimicrobial Therapy in Haematologic Patients With Febrile Neutropenia
Brief Title: Study to Reduce Duration of Antibiotic Therapy in Haematological Patients With Fever and Neutropenia
Acronym: HOWLONG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2011-005152-34
Record Dates: First submitted 2012-04-17; First posted 2012-04-20 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Febrile Neutropenia
Keywords: febrile neutropenia; antimicrobial treatment; procalcitonin
MeSH Terms: conditions — Febrile Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Arm (Experimental): Empirical antimicrobial treatment discontinuation
  Interventions: Drug: Empirical antimicrobial treatment discontinuation
- Control Arm (Active Comparator): Standard empirical antimicrobial treatment discontinuation
  Interventions: Drug: Standard empirical antimicrobial treatment discontinuation

INTERVENTIONS:
Drug: Empirical antimicrobial treatment discontinuation — Empirical antimicrobial treatment discontinuation will occur when the patient is: Afebrile, with resolution of signs, symptoms and test abnormalities secondary to complementary source of infection and with normalization of vital signs for ≥ 72 h.
  Other Names: Clinical rules for finalization of antimicrobial therapy
  Arms: Experimental Arm
Drug: Standard empirical antimicrobial treatment discontinuation — The empirical antimicrobial treatment discontinuation will occur when the patient is:
  The neutrophil count is above 500 million per mm3.
  Other Names: Laboratory rules for finalization of antimicrobial therapy
  Arms: Control Arm

SUMMARY:
Clinical trial intended to reduce the antibiotic therapy duration in "in-hospital" patients with haematological diseases who develop fever and low white blood cell count (neutropenia).

DETAILED DESCRIPTION:
The optimal duration of the empirical antimicrobial therapy (AT) in hematological patients with febrile neutropenia (FN) is unknown. The Infectious Diseases Society of America (IDSA) recommends maintaining AT at least until the neutropenia is recovered, because literally "years of experience have proven this approach to be safe and effective". This recommendation is likely to cause unnecessarily prolonged treatments, and is against the urgent need of optimizing the antimicrobial therapy proposed by IDSA. The main objective of this study is to establish whether an individualized clinical protocol is better than the standard criteria (recovery of neutropenia as the criterion to suspend the empirical AT in hematological patients with FN).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (equal or older than 18 years) of both sexes admitted in the Department of Clinical Hematology who develop a febrile neutropenia. Including fever with unknown source and fever secondary to infection focus of clinical diagnosis without laboratory confirmation.
* Informed consent signed.

Exclusion Criteria:

* Fever with etiologic diagnosis.
* Patients with epilepsy.
* Pregnant or lactating women.
* Patients with HIV infection.
* Patients with severe renal failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2012-04; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of days on which patient is free of antimicrobial treatment | 28 days following the initiation of empiric antibiotic treatment.
  Protocol visits: Screening visit, Randomization visit, at 72h. of apyrexy (visit 1), at clinical recovery (visit 2), at recovery of neutropenia (visit 3), at relapsing fever (visit 4) and at 28 days (final visit).

SECONDARY OUTCOMES:
Crude mortality | 28 days following the initiation of empiric antibiotic treatment.
  Number of died patients
Number of days of fever | 28 days following the initiation of empiric antibiotic treatment
  Number of days of fever

CONTACTS AND LOCATIONS:
Overall Officials: José M Cisneros Herreros, PhD, Study Director — Virgen del Rocío University Hospital/ Biomedicine Institute of Seville (IBIS)
Locations (6):
- Spain (6):
  - Hospital de Jerez, Jerez de la Frontera, Cádiz
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clínic, Barcelona
  - Bellvitge University Hospital, Barcelona
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Virgen del Rocío University Hospital, Seville

REFERENCES:
- [Derived] Aguilar-Guisado M, Espigado I, Martin-Pena A, Gudiol C, Royo-Cebrecos C, Falantes J, Vazquez-Lopez L, Montero MI, Rosso-Fernandez C, de la Luz Martino M, Parody R, Gonzalez-Campos J, Garzon-Lopez S, Calderon-Cabrera C, Barba P, Rodriguez N, Rovira M, Montero-Mateos E, Carratala J, Perez-Simon JA, Cisneros JM. Optimisation of empirical antimicrobial therapy in patients with haematological malignancies and febrile neutropenia (How Long study): an open-label, randomised, controlled phase 4 trial. Lancet Haematol. 2017 Dec;4(12):e573-e583. doi: 10.1016/S2352-3026(17)30211-9. Epub 2017 Nov 15. PMID 29153975

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2015-02-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT01581333/Prot_ICF_000.pdf